CLINICAL TRIAL: NCT04924361
Title: Exploring Biomarkers in Age Stratified PUMCH Dementia Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, gaojing, Professor, Department of Neurology, Peking Union Medical College Hospital
Other Study IDs: PUMCH Dementia Cohort Research
Record Dates: First submitted 2021-05-18; First posted 2021-06-14 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Dementia; Dementia, Vascular; Dementia Frontal; Dementia, Mixed; Dementia Alzheimers; Dementia With Lewy Bodies
Keywords: Biomarkers; Diagnosis
MeSH Terms: conditions — Dementia; Dementia, Vascular; Mixed Dementias; Alzheimer Disease; Lewy Body Disease; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early onset dementia: Dementia patients with onset age lower than 65y/o
- Late onset dementia: Dementia patients with onset age between 65y/o and 85y/o
- Oldest old dementia: Dementia patients with onset age older than 85y/o
- Cognitive normal control: cognitive normal control

SUMMARY:
Biomarkers are important for early and precise diagnosis of dementia. However, the causes of dementia in different age are different. We designed an age stratified dementia cohort and tried to explore biomarkers of different groups of dementia, incorporating neuropsychology, multi-model neuroimaging, metabolics and proteomics based fluid biomarkers as well as genetic biomarkers. Autopsy after clinical follow up help to verify the biomarkers.

DETAILED DESCRIPTION:
Baseline data collection and cohort establishing: Detailed clinical information including demographic data, clinical history, past history and physical examination are collected. Formatted neuropsychological battery is used in all patients, including screening tests (MMSE, MoCA-PUMCH, ADL, HAD) and domain specific evaluation (Memory, executive function, visual spatial, calculation, language). Samples including serum, CSF, urine, skin, saliva are stored. Every patient is followed up every 6 months. Autopsy brain tissue will be collected if patients died.

Multi-model neuroimaging evaluation: Structure and functional brain 3T-MRI; 7T-MRI； PET-CT including FDG, Aβ（18F-AV45）,tau（18F-THK5317, 18F-T807）; EEG

Multi-omics biomarkers research:

CSF AD biomarkers (Aβ40,42, ptau181, ttau, NfL, Neurogranin), comparison of different methods, including ELISA, Electrochemical, Mass Spectroscopy. The standardization of CSF biomarkers analysis in China.

Exploring new fluid biomarkers: CSF and Urine proteomics; CSF and serum glycomics and metabolomics. To explore new biomarkers in differentiation of different causes of dementia, age onset and prognosis of dementia.

Genetic biomarkers evaluation: including pathogenic gene mutation panel examination and WES.

Data analysis and biomarkers evaluation: Dementia patients are stratified based on age onset, cause of dementia, cognition severity, effect of therapy, prognosis. Identify multi-omics biomarkers in different groups. Comparing the relationships between biomarkers and clinical presentations as well as neuroimaging. Autopsy based accurate diagnosis help further defining biomarkers.

Acquiring stratified biomarkers with high sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Neurodegenerative dementia diagnosis based on 2011 NIA-AA criteria of Dementia
* Fixed care giver and can follow up regularly

Exclusion Criteria:

* Not demented, including MCI
* Systemic severe diseases and severe vision or hearing problem effecting follow up and neuropsychological evaluation
* Without fixed care giver
* Reject informed consent
* Expected life shorter than 2 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We included age stratified dementia (early onset, late onset, oldest old) , including AD, FTD,VaD, DLB and mixed dementia. Also we include cognitive normal controls.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Incorporating age stratified biomarkers into the diagnosis of dementia | Through study completion,an average of 5 years
  Comparing the relationships between biomarkers and clinical presentations as well as neuroimaging. Incorporate biomarkers into the accurate and early diagnosis of dementia

SECONDARY OUTCOMES:
Establishing dementia cohort including detailed clinical information, fluid samples and brain bank | Through study completion,an average of 5 years
  Detailed clinical information including demographic data, clinical history, past history and physical examination are collected. Formatted neuropsychological battery is used in all patients, including screening tests (MMSE, MoCA-PUMCH, ADL, HAD) and domain specific evaluation (Memory, executive function, visual spatial, calculation, language). Samples including serum, CSF, urine, skin, saliva are stored. Every patient is followed up every 6 months. Autopsy brain tissue will be collected if patients died after informed consent.
Exploring 5-10 kinds of age stratified biomarkers, including neuropsychology, neuroimaging, fluid biomarkers and genetic biomarkers | Through study completion,an average of 5 years
  Find out age stratified biomarkers with high sensitivity and specificity, including neuropsychology, Multi-model neuroimaging, Multi-omics fluid biomarkers and genetic biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Jing Gao, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuruppu DK, Matthews BR. Young-onset dementia. Semin Neurol. 2013 Sep;33(4):365-85. doi: 10.1055/s-0033-1359320. Epub 2013 Nov 14. PMID 24234358
- [Background] Rabinovici GD. Late-onset Alzheimer Disease. Continuum (Minneap Minn). 2019 Feb;25(1):14-33. doi: 10.1212/CON.0000000000000700. PMID 30707185
- [Background] Yang Z, Slavin MJ, Sachdev PS. Dementia in the oldest old. Nat Rev Neurol. 2013 Jul;9(7):382-93. doi: 10.1038/nrneurol.2013.105. Epub 2013 Jun 4. PMID 23732531
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606